CLINICAL TRIAL: NCT07162493
Title: Attachment and Child Health (ATTACH) Added to Treatment As Usual Versus Treatment As Usual Alone for Parents With Psychosocial Problems: A Feasibility Randomized Controlled Trial
Brief Title: ATTACH in Denmark: A Feasibility Randomized Controlled Trial
Acronym: AiD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johanne Smith-Nielsen (Other)
Collaborators: University of Calgary Cumming School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Johanne Smith-Nielsen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AID-RCT-2025
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Mentalization; Recruitment of Participants; Adherence, Treatment; Drop Out; Parenting Intervention; Vulnerable Families; Feasibility Studies
Keywords: parenting; mentalizing; intervention; feasibility
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Between-subjects design with 1 factor (intervention type) and 2 levels: (a) ATTACH™ + Treatment As Usual and (b) Treatment As Usual alone. Participants are randomized 1:1 using stratified block randomization (municipality, child sex).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATTACH(TM) parenting program added to treatment as usual (Experimental): Developed in Canada by Professor Nicole Letourneau and Dr. Martha Hart, the Attachment and Child Health (ATTACH) parenting program is an intervention for parents of children aged 0-5 years, aiming at improving parental mentalizing skills. It is a manualized, short-term intervention consisting of 10 sessions. Although it can function as a stand-alone intervention, ATTACH has been developed and tested as an add-on to existing practices. Thus, in this trial, the experimental intervention will be ATTACH added to Treatment As Usual.
  Interventions: Behavioral: ATTACH; Behavioral: Treatment as Usual (TAU)
- Treatment as usual (Active Comparator): The control intervention is Treatment As Usual (TAU) provided at the specific trial site, which consists of the standard services and support typically offered to families by the local social- and healthcare systems within municipalities.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: ATTACH — ATTACH(TM) is a manualized, 10-session, mentalizing/reflective functioning-based parenting program, with one 45-60-minute weekly session. It is conducted individually with one parent focusing on one child throughout the program; however, a co-parent/parental support person will participate in session 7 and session 9. A session includes three components to facilitate parental reflective functioning: 1)Video-review of parent-child interaction, 2) reflection on a hypothetical situation (pre-defined for each session), and 3) reflection on a mildly stressful situation from the parent's everyday life with the child. The parent's reflective process is supported by handouts, e.g., "emotion cards". All material used in the sessions have been translated into Danish, and the wording have been modified to fit with the cultural context, based on feedback from two pilot studies. ATTACH is facilitated by professionals employed at the family centers, who have been trained and certified in ATTACH.
  Arms: ATTACH(TM) parenting program added to treatment as usual
Behavioral: Treatment as Usual (TAU) — Treatment As Usual (TAU) consists of the standard services and support typically offered to families by the local social- and healthcare systems within each municipality. These services vary depending on individual needs, risk assessment of the family, and municipal practices, but often include individual and/or group-based parenting support or therapeutic services at the trial site and/or in the parent's home. TAU may also involve referrals to additional resources or interventions deemed necessary by social authorities or healthcare providers (e.g., psychiatric treatment in the region). The control group will not receive the ATTACH™ program but will have access to all relevant standard care options available within their municipality. TAU can be delivered by different professionals, such as health visitors, social workers, family therapists/counsellors or clinical psychologists. For more details on TAU services at each trial site, see the attached project protocol.

SUMMARY:
The goal of this feasibility randomized controlled pilot trial is to learn whether the trial can be done as planned, and to investigate if the 10-session parenting program "ATTACH(TM) increases mentalizing skills (the ability to reflect on thoughts and feelings) in parents of children between 0-5 years of age, who are receiving support for psychosocial problems in their municipal family treatment center.

The main questions the trial aims to answer are:

* How many eligible parents agree to participate in the random allocation to treatment?
* How many parents allocated to receive "ATTACH(TM) will have completed the program 5 months after allocation (at least 7 out of 10 sessions)?
* How many parents complete the data collection 5 months after allocation on the primary exploratory clinical outcome, i.e., parental mentalizing skills?
* Do parents who received the ATTACH(TM) program show more increase in their mentalizing skills, compared to parents, who did not receive treatment with ATTACH(TM)?

Researchers will compare ATTACH, added to Treatment as Usual, with Treatment as Usual without ATTACH in three municipal family treatment centers located in the Capital Region of Denmark.

Participants will:

1. Take part in baseline data collection with a survey, video observation of parent-child interaction, and an interview assessing mentalizing skills.
2. Be randomly allocated to receive treatment in their local family center with or without ATTACH.
3. Take part in data collection 5 months after being allocated to either group, as well as participate in an interview about their experiences with the treatment they received.
4. After one year, the research group will follow up on the current treatment/support needs of the families, who were allocated to either group.

DETAILED DESCRIPTION:
See the attached project protocol for a detailed description

ELIGIBILITY:
Inclusion criteria

* Child aged 0 - 5.7 years at enrollment.
* Speaks Danish or English sufficiently to take part in assessments and intervention without an interpreter.
* Both parents provide consent in case of shared child custody. Parents experience psycho-social problems that have resulted in referral to the family treatment center on the basis of legislation from the Danish Child Act ("Barnets Lov"), under the following Sections defining support needs: Section 29: Family counselling: Includes open access to family counselling as an early preventive effort. In this context, the counselling may involve referring the family to other departments within the municipality or to other relevant authorities that can provide the appropriate guidance and support. Section 30: Early preventive intervention: Includes a variety of approaches, such as consultancy services and participation in network or discussion groups to address and prevent challenges faced by the family at an early stage. Section 32: Supportive interventions: May be initiated on the basis of a preliminary assessment or a child welfare investigation pursuant to Sections 19 and 20 of the Child Act, or concurrently with the completion of such an assessment or investigation. Support may include practical, pedagogical, or other types of support in the home; appointment of a permanent contact person for the entire family; family therapy or individual treatment for the child or young person; family placement involving residential care in a foster family, an approved child and youth residential facility, or a housing facility; supportive placement in a foster family or in an approved child and youth residential facility; other forms of assistance aimed at providing counseling, treatment, and practical and pedagogical support.
* Parents who have their child in out-of-home placement /foster care (with or without consent).
* Parental psychosocial problems such as (but are not limited to) mental health problems, cognitive difficulties, substance abuse, poverty, social isolation, adverse childhood experiences, functional or somatic disorders, criminal involvement, domestic violence, having a child with emotional regulation difficulties, having a child with developmental problems, having a child with functional or somatic problems, having a child with internalizing or externalizing problems.

Exclusion Criteria:

* Child is older than 5.7 years at enrollment.
* Parent does not speak Danish or English sufficiently to take part in assessments and intervention without an interpreter.
* Consent cannot be obtained from both parents in case of shared child custody.
* The parent is known to move to a different municipality within 5 months from randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcomes | We will assess the proportion of three criteria at 5 months after randomization in both arms.
  As this is a feasibility trial, the primary aim is to assess feasibility rather than efficacy. We have therefore pre-defined three criteria that will guide our evaluation of whether a future large-scale trial is feasible:
  1. Inclusion proportion: At least 25% of eligible parents consent to participation and randomization.
  2. Compliance proportion: At least 50% of parents randomized to the ATTACH group complete ≥7 of 10 sessions.
  3. Completion proportion: At least 70% of randomized participants provide complete data on the primary clinical exploratory outcome at 5 months.
Primary clinical exploratory outcome - parental mentalizing/insightfulness | IA is assessed at baseline prior to randomization and again at 5 months post randomization.
  Parents are assessed for their mentalizing capacity using the Parental Insightfulness Assessment interview (IA). Parental insightfulness is defined as the capacity to see things from the child's point of view. The IA is conducted as follows: 1) Video recordings of parent and child interacting. 2) Reviewing 2x2 minute video segments with the parent while conducting the interview. 3) transcription and coding of interview. The interview procedure has been modified to be in accordance with the trial's videorecording procedures, which originally includes reviewing of three video segments, while for this trial, we will include two video segments. The IA consists of 10 different scales, each given a score on a 9-point scale (low to high). Based on the scale scores, the parent is classified into one of four categories: Positively Insightful; One-sided; Disengaged; or Mixed. However, for this study, we will use scale scores from 1 to 9 as the primary indication of parental mentalizing capacity

SECONDARY OUTCOMES:
Parental Reflective Functioning | Assessed at baseline prior to randomization and at 5 months post randomization
  Parental reflective functioning will be assessed using the Parental Reflective Functioning Questionnaire (PRFQ) for parents of children from 1 to 5 years, while the infant version (PRFQ-I) is used for children aged 0-1 year. The PRFQ/I is a self-report questionnaire consisting of 18 and 15 items, respectively. Item are scored on a 7-point Likert scale, ranging from 1 (completely disagree) to 7 (completely agree). Each item corresponds to one of three subscales reflecting aspects of parental reflective functioning, i.e., Interest and Curiosity in the child's thoughts and feelings; Certainty about the child's mental states; and pre-mentalizing (a non-mentalizing stance). The PRFQ/I is included in an online survey.
Reflective functioning, general | Assessed at baseline prior to randomization and at 5 months post randomization
  To assess non-parenting specific reflective functioning, we will use the 8-item version of the Reflective Functioning Questionnaire (RFQ-8). Each item of the RFQ-8 is scored on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The RFQ-8 is included in an online survey
Parental Mind-Mindedness | Assessed at baseline prior to randomization and at 5 months post randomization
  Mind-Mindedness (MM) reflects the parent's tendency to treat the child as a psychological individual in term of how they describe their child from a mentalizing stance, i.e., the child's thoughts, feelings, intentions etc. We will use the representational measure of MM, using parental written descriptions of their child: In the beginning of the online survey, the parent is probed to "describe your child", which will be coded according to the standard procedures. The MM is included in an online survey
Parent-child interaction quality, free-play | Assessed at baseline prior to randomization and at 5 months post randomization
  At the home-visit, a trial investigator instructs the parent to play with their child as they normally would for a total duration of seven minutes. If the child is seven months or older, the interaction includes a mild frustration episode after three minutes, lasting for one minute (parent is instructed to remove child's preferred toy and keep it away from child for one minute). This will be assessed using the method Coding Interactive Behavior, assessing mainly parental sensitivity. The CIB consist of 33 items, 18 related to parental behavior (e.g., acknowledging child signals); eight to the child's behavior (e.g., initiation), and five to the dyad (e.g., dyadic reciprocity), and, finally, two scales are on the lead-lag of the interaction (i.e., child- or parent-led). All items are rated on a scale ranging from 1 (representing the minimal level of the behavior) to 5 (representing the highest level), with the possibility of providing half points.
Parent-child interaction quality, teaching situation | Assessed at baseline prior to randomization and at 5 months post randomization
  At the home visit, the trail investigator instructs the parent to pick a task from a pre-defined list, that they would like to teach their child (e.g., stack blocks or draw a circle on paper). The recording cannot be shorter than 2 minutes and no longer than 5 minutes. This will be coded using the Parent-Child Interaction Teaching Scale (PCITS). The PCITS is made up of 73 binary items organized into six subscales, four pertaining to the parent and two to the child: Caregiver's Sensitivity to Cues; Caregiver's Response to the Child's Distress; Caregiver's Social-Emotional Growth Fostering; Caregiver's Cognitive Growth Fostering; Child's Clarity of Cues; and, Child's Responsiveness to Caregiver. Each item is scored either "yes" or "no", depending on if the described behavior is present during the teaching episode.
Child development | Assessed at baseline prior to randomization and again at 5 months post randomization
  We will use the Ages and Stages Questionnaire, 3rd edition (ASQ-3) to evaluate child global development. It consists of 30 items corresponding to different subscales of developmental domains, i.e., cognitive skills (communication, problem-solving, and personal-social) and motor skills (gross and fine). The ASQ-3 identifies children at risk for adverse mental health and development. While the ASQ-3 is developed as a self-report questionnaire, it will be administered by an investigator together with the parent and child at the data collection visit to strengthen validity of responses.
Child externalizing and internalizing problems and wellbeing | Assessed at baseline prior to randomization and at 5 months post randomization
  This will be assessed using the Child Behavior Checklist (CBCL) for Children Aged 1.5-5 years. The CBCL measures internalizing and externalizing problems as well as sleep difficulties and somatic problems. The CBCL consist of 99 items, each scored on a 3-point scale from 0=not true, 1=somewhat or sometimes true, 2=very true or often true), with higher scores indicating more dysfunction and problems. The CBCL is included in an online survey.
Parental depression | Assessed at baseline prior to randomization and at 5 months post randomization
  To assess parental depression we will use the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item self-report questionnaire, with each item scored from 0-3 (range 0-30). It is designed to screen for possible depression based on how the parent has been feeling within the past 7 days, with higher scores indicating higher levels of depressive mood. The EPDS is included in the online survey.
Parenting stress | Assessed at baseline prior to randomization and at 5 months post randomization
  We will use the Parenting Stress Index Fourth Edition short Form (PSI-4-SF), which is a 36-item self-report questionnaire assessing parenting stress on three domains: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, as well as a Total Stress score, with higher scores indicating higher parenting stress. Each item is scored on a 5-point Likert scale (from Strongly Agree to Strongly Disagree). Clinically significant cut-offs have been established. The PSI-4-SF is included in the online survey.
Resilience and coping with stress | Assessed at baseline prior to randomization and at 5 months post randomization
  This will be assess by the Brief Resilience Scale (BRS), which consists of six items scored on a 5-point Likert Scale (from Strongly Disagree to Strongly Agree, range 6-30), with higher scores indicating more resilience and increased ability to bounce back from stress. The BRS is included in the online survey
Family functioning | Assessed at baseline prior to randomization and at 5 months post randomization
  To assess overall healthy functioning or dysfunction of intrafamilial relationships We will use the McMaster Family Assessment Device - Short Version (FAD). It is a 12 item self-report questionnaire, with each item scored on a 4-point Likert Scale ranging (from Completely Disagree to Completely Agree), with higher scores indicative of more dysfunction. The FAD is included in the online survey

OTHER OUTCOMES:
Support needs of family one year after randomization | Assessed one year post randomization
  One year after randomization, we will retrieve information from the family treatment units on the current support needs of the family. This is to assess whether the family has required additional or ongoing support, or whether their need for support has changed.

CONTACTS AND LOCATIONS:
Overall Officials: Johanne Smith-Nielsen, PhD, associate professor, Principal Investigator — Centre of Excellence in Early Intervention and Family Studies, Department of Psychology, University of Copenhagen; Katrine Isabella Wendelboe, PhD, Principal Investigator — Centre of Excellence in Early Intervention and Family Studies, Department of Psychology, University of Copenhagen; Nicole Letourneau, PhD, professor, Principal Investigator — Faculty of Nursing and Cumming School of Medicine, University of Calgary
Locations (3):
- Denmark (3):
  - Center for Sociale Indsatser, Gribskov
  - Poppelgården Familiecenter, Hvidovre
  - Familie- og Dagtilbudscenter, Høje Taastrup

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because our dataset involves subjects who will not explicitly consent to the publication of their pseudonymized data which is required to comply with the Danish Data Protection Act. Therefore, publishing the dataset does not align with the ethical standards of data management and regulations upheld at the University of Copenhagen. Data are available from the Data Management and Information Security department at the Department of Psychology, University of Copenhagen (contact via legal@samf.ku.dk) for researchers who meet the criteria for access to confidential data.

REFERENCES:
- See also: Related Info — https://psy.ku.dk/cif/english/research/attach-in-dk/